CLINICAL TRIAL: NCT04731779
Title: Cannabidiol and Autonomic Function in Individuals at Rest
Brief Title: Cannabidiol and Autonomic Function at Rest
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Castleton University (Other)
Responsible Party: Principal Investigator, Andrea Corcoran, Assistant Professor of Exercise Science, Castleton University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: VRBN Pilot 2021_Corcoran
Record Dates: First submitted 2021-01-21; First posted 2021-02-01 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Each participant will receive a different dose in consecutive weeks (4 doses total, one of which is a placebo), thus serving as their own control.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will ingest 3ml of non-CBD containing MCT (medium-chain triglycerides) oil.
  Interventions: Drug: Placebo
- 25 mg (Experimental): Participants will ingest 3ml of MCT (medium-chain triglycerides) oil containing 25 mg of CBD.
  Interventions: Drug: cannabidiol
- 50 mg (Experimental): Participants will ingest 3ml of MCT (medium-chain triglycerides) oil containing 50 mg of CBD.
  Interventions: Drug: cannabidiol
- 200 mg (Experimental): Participants will ingest 3ml of MCT (medium-chain triglycerides) oil containing 200 mg of CBD.
  Interventions: Drug: cannabidiol

INTERVENTIONS:
Drug: cannabidiol — Cannabidiol oral product formulated in MCT (medium chain triglyceride) oil
  Other Names: CBD
  Arms: 200 mg; 25 mg; 50 mg
Drug: Placebo — Placebo oral product formulated in MCT (medium chain triglyceride) oil
  Arms: Placebo

SUMMARY:
Cannabidiol (CBD) is one of 700 chemicals derived from the Cannabis sativa plant and is both legal and widespread for distribution in the state of Vermont. The central hypothesis of this proposal is that in apparently healthy adults, acute CBD favorably affects the autonomic nervous system and that this will be evident by an increase in heart rate variability. The overall goal is to understand how CBD affects the autonomic and cardiovascular systems at rest, and when perturbed. The investigators will study a narrow age range of adults, administer varying acute doses of CBD, characterize baseline cardiovascular variables, and record responses to autonomic challenge maneuvers. This will provide the framework to assess potential therapies and/or risk factors of CBD, particularly as it relates to healthy individuals. More information that is so widely taken, especially one that targets receptors known to be involved in cardiovascular signaling pathways is imperative.

DETAILED DESCRIPTION:
The study will be conducted in the Exercise Physiology Laboratory in the Jeffords Science Building at Castleton University. Participants will be asked to fast overnight, avoid beverages or food containing caffeine, alcohol, or CBD for at least 12h, and to not perform physical effort for 6h prior to each session.

During the initial session, individuals will: have their height and body mass measured, complete a health history questionnaire, and sign a consent form approved by Castleton University's Institutional Review Board. Prior to data collection, individuals will be advised of the possible risks, methods, and potential benefits of this study. They will also be familiarized with the noninvasive cardiovascular monitoring equipment, which they will be putting on themselves. These include an automated blood pressure (BP) cuff and a heart rate (HR) chest strap monitor.

On the day of each experiment, participants will be given a standardized meal and asked to put on the BP cuff and HR monitor. Individuals will remain seated for the length of the experiment (doing nothing or reading). Baseline measurements will be taken remotely following 15 minutes of rest. Under supervision, participants will be asked to consume oral CBD oil (0mg, 25 mg, 50 mg, or 200mg), infused in non-CBD containing MCT (medium-chain triglycerides) oil to standardize dose volume of 3ml. Assessments will be measured remotely at intervals up to 2.5 hours after ingestion. The study will be double-blind, thus neither the participant nor researcher will be aware of the CBD dose for a particular session. Participants will be asked to return for 3 additional consecutive weeks, each session will be a different dose of CBD.

In the final experimental session (to be completed after initial analyses of dose responses), participants will be given a standardized meal and asked to put on the blood pressure cuff and HR monitors. Individuals will remain seated for the length of the experiment. Following 15 minutes of rest, participants will be asked to perform two autonomic stress tests: the isometric hand grip test, and the cold face test. First, the maximum voluntary contraction (MVC) for the isometric hand grip test will be assessed. Participants will be asked to press a handgrip dynamometer with full strength. To perform the isometric handgrip test, participants will again use the dynamometer and maintain handgrip at 30 percent MVC for 2 min. A recovery period of 10 minutes between each test will be observed. For the cold face test, a cold compress (1-2 degrees Celcius) will be applied to the forehead and maxillary region of the subjections face for 2 min. Following these baseline tests, participants will be asked to consume a dose of CBD (determined following analyses of the initial 4 sessions) and perform the two autonomic stress tests again 2h post ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-35 years of age.
* Participants must agree to fast and abstain from food or beverages containing alcohol, caffeine, or CBD for 12 hours prior to each experimental session.
* Completion of Health History Questionnaire with report indicating overall good health.
* The ability to comprehend and satisfactorily comply with protocol requirements.
* Written informed consent given prior to beginning the study.

Exclusion Criteria:

* Current medications that might influence the cardiovascular and/or autonomic systems.
* Women who are pregnant or lactating.
* Participants who have a history of adverse reactions to cannabidiol will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) as assessed by time-domain analysis: standard deviation of RR intervals. | 4 weeks
  Time-domain measurements quantify the amount of variability of the heart's interbeat (RR) intervals and include the metric: standard deviation of RR intervals (SDNN). Higher values indicate greater HRV.
Change in heart rate variability (HRV) as assessed by time-domain analysis: root mean square of successive differences. | 4 weeks
  Time-domain measurements quantify the amount of variability of the heart's interbeat (RR) intervals and include the metric: root mean square of successive differences (RMSSD). Higher values indicate greater HRV.
Change in heart rate variability (HRV) as assessed by frequency-domain analysis: high-frequency (HF). | 4 weeks
  Frequency-domain measurements estimate the distribution of absolute or relative power into four heart rate oscillation frequency bands: ultra-low-frequency (ULF), very-low-frequency (VLF), low-frequency (LF) and high-frequency (HF). A high HF reflects parasympathetic dominance.
Change in heart rate variability (HRV) as assessed by frequency-domain analysis: low-frequency (LF). | 4 weeks
  Frequency-domain measurements estimate the distribution of absolute or relative power into four heart rate oscillation frequency bands: ultra-low-frequency (ULF), very-low-frequency (VLF), low-frequency (LF) and high-frequency (HF). LF reflects both sympathetic and parasympathetic activity.
Change in heart rate variability (HRV) as assessed by frequency-domain analysis: LF/HF ratio. | 4 weeks
  A low LF/HF ratio reflects parasympathetic dominance, whereas a high LF/HF ratio reflects sympathetic dominance.
Change in magnitude of autonomic stress test responses as assessed by changes in blood pressure. | 1 day
  Responses to autonomic stress test include a change in blood pressure if sympathetic outflow is activated. The magnitude of change will be compared before and after CBD ingestion.
Change in magnitude of autonomic stress test responses as assessed by changes in heart rate. | 1 day
  Responses to autonomic stress test include a change in heart rate if parasympathetic outflow is activated. The magnitude of change will be compared before and after CBD ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Castleton University, Jeffords Science Building, Castleton, Vermont, United States

IPD SHARING:
Plan to Share IPD: No